CLINICAL TRIAL: NCT02774226
Title: Long Term Nitric Oxide Bioavailability on Vascular Health in Chronic Obstructive Pulmonary Disease
Acronym: COPD-LT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ryan Harris, Principal Investigator, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COPD-LT
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Flow-Mediated Dilation; Kuvan; Antioxidant; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — sapropterin; Ascorbic Acid; Vitamin E; Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetrahydrobiopterin (BH4) (Experimental): Blood samples, flow-mediated dilation, arterial stiffness, lung function, and microvascular function will be performed at baseline and 12 weeks following 5mg/kg of Kuvan® or sapropterin dihydrochloride which is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4), taken once a day.
  Interventions: Drug: Tetrahydrobiopterin (BH4)
- Antioxidant Cocktail (Experimental): Blood samples, flow-mediated dilation, arterial stiffness, lung function, and microvascular function will be performed at baseline and 12 weeks following an anti-oxidant cocktail (vitamin C 1000 mg, vitamin E 400 IU, and alpha lipoic acid 600 mg) taken once a day.
  Interventions: Dietary Supplement: Antioxidant Cocktail

INTERVENTIONS:
Drug: Tetrahydrobiopterin (BH4) — 12 week intervention
  Other Names: Kuvan (Sapropterin Dihydrochloride)
  Arms: Tetrahydrobiopterin (BH4)
Dietary Supplement: Antioxidant Cocktail — 12 week intervention
  Other Names: Vitamin C; Vitamin E; Alpha Lipoic Acid
  Arms: Antioxidant Cocktail

SUMMARY:
Chronic obstructive pulmonary disease (COPD) affects up to 14 million people and is among the top five leading causes of death worldwide. Although COPD is a disease of the lungs, recent evidence indicates that COPD is associated with multiple systemic consequences including vascular endothelial dysfunction. Recently, it has been suggested that more patients with COPD die from cardiovascular disease and coronary heart disease than of direct pulmonary complications. Examination of the mechanisms that contribute to a reduction nitric oxide (NO) bioavailability resulting in vascular endothelial dysfunction in patients with COPD are important as endothelial dysfunction has been indicated to be an independent predictor of future atherosclerotic cardiovascular disease and events.

DETAILED DESCRIPTION:
Researchers have found a link between chronic obstructive pulmonary disease (COPD) and heart disease; however, a link is all they have found. In a previously funded grant, using a double blind, randomized experimental design, the investigators explored the effect of an acute dose of Kuvan or an antioxidant cocktail (1000mg of vitamin C, 600IU of vitamin E, and 600mg alpha-lipoic acid) on vascular health in patients with COPD. Consequently, the investigators found in separate experiments, that a single dose of both antioxidants and Kuvan transiently improves vascular health in patients with COPD. The current project is an attempt to expand on the investigator's previous findings and explore the effects of sub-chronic use of antioxidants and Kuvan on sustaining the improvements in vascular health in COPD.

ELIGIBILITY:
Inclusion Criteria:

* patients with medically diagnosed COPD
* apparently healthy controls

Exclusion Criteria:

* FEV1/FVC >0.7 (normal lung function in patients only)
* Clinical diagnosis of heart disease or diabetes
* Vasoactive medications (i.e. nitrates, beta-blockers, Viagra etc.)
* uncontrolled high blood pressure
* high blood pressure in your lungs
* thyroid problems
* Fluid in the lungs
* Sleep apnea
* Anemia
* Raynaud's Phenomenon
* GI bleeding
* Gangrene of the digits
* History of low platelets or coagulopathies
* Phenylketonuria (PKU)
* Any allergy to Kuvan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, Ph.D, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Tetrahydrobiopterin (BH4): Blood samples, flow-mediated dilation, arterial stiffness, lung function, and microvascular function will be performed at baseline, 4 weeks, 8 weeks, and 12 weeks following, 5mg/kg, 10mg/kg, or 20mg/kg of Kuvan® or sapropterin dihydrochloride which is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4), taken once a day.
  Tetrahydrobiopterin (BH4): 12 week intervention
- Antioxidant Cocktail: Blood samples, flow-mediated dilation, arterial stiffness, lung function, and microvascular function will be performed at baseline, 4 weeks, 8 weeks, and 12 weeks following an anti-oxidant cocktail (vitamin C 1000 mg, vitamin E 400 IU, and alpha lipoic acid 600 mg) taken once a day.
  Antioxidant Cocktail: 12 week intervention
Period: Overall Study
Arm/Group | Tetrahydrobiopterin (BH4) | Antioxidant Cocktail
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tetrahydrobiopterin (BH4) | Antioxidant Cocktail | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (5) | 57 (6) | 59 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow Mediated Dilation
Description: Brachial artery FMD induced by reactive hyperemia assessed vascular endothelial function at baseline and 12 weeks after treatment.
Time Frame: Change from Baseline and 12 weeks
Population: Data was not usable on one participant in the antioxidant group. Too much artifact.
Measure: Mean (Standard Deviation); unit: percentage of flow mediated dilation
Arm/Group | Tetrahydrobiopterin (BH4) | Antioxidant Cocktail
Number analyzed (Participants) | 8 | 6
percentage of flow mediated dilation | 0.26 (2.57) | -1.5 (3.86)

2. Secondary Outcome: Change in PWV (Pulse Wave Velocity)
Description: Change in pulse wave velocity (carotid to femoral) as measured using tonometry with the Sphygmocor Xcel system at baseline and after 12 weeks of treatment.
Time Frame: Change from Baseline and 12 weeks
Population: Unable to obtain pulse wave on 2 participants in the AOX group.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Tetrahydrobiopterin (BH4) | Antioxidant Cocktail
Number analyzed (Participants) | 8 | 5
m/s | -0.36 (0.66) | 0.34 (0.86)

3. Secondary Outcome: FEV1 %Predicted
Description: Forced Expiratory Volume in 1 second. Pulmonary Function Test (PFT).
Time Frame: Change from Baseline and 12 weeks
Population: Unable to obtain valid lung function on one participant in the BH4 group as well as one participant in the AOX group.
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Tetrahydrobiopterin (BH4) | Antioxidant Cocktail
Number analyzed (Participants) | 7 | 6
percentage of predicted | -3.6 (6.3) | -4.2 (10.9)

4. Secondary Outcome: Percent of ACH to Heat Max
Description: The laser imaging camera is a special camera that shines a low energy laser light on the surface of the skin to measure blood flow. The FLPI makes graphs, photos, and movies of skin blood flow. Acetylcholine is a vasoactive substance that will be used to increase skin blood flow. This variable is the percent of dilation caused by acetylcholine out of the max dilation cause by the warm water bath (44 C).
Time Frame: Change from Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Tetrahydrobiopterin (BH4) | Antioxidant Cocktail
Number analyzed (Participants) | 8 | 7
percent | 4.2 (15) | -0.8 (41.6)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Tetrahydrobiopterin (BH4) | Antioxidant Cocktail
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02774226/Prot_SAP_000.pdf